CLINICAL TRIAL: NCT07236411
Title: A Randomized, Double-blind, Phase 1 Study to Evaluate the Absolute Bioavailability of Cizutamig Following Single Intravenous or Subcutaneous Administration in Healthy Adult Participants
Brief Title: Absolute Bioavailability Study of Cizutamig in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Candid Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CND106-001
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants Study
Keywords: healthy volunteer; pharmacokinetics; pharmacodynamics; immune system; cizutamig; T cell engager; bioavailability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SC injection of cizutamig (Experimental): cizutamig subcutaneous injection
  Interventions: Biological: cizutamig
- SC injection of placebo (Placebo Comparator): placebo subcutaneous injection
  Interventions: Other: Placebo
- IV infusion of cizutamig (Experimental): IV cizutamig
  Interventions: Biological: cizutamig
- IV infusion of placebo (Placebo Comparator): IV placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: cizutamig — cizutamig will be dosed SC or IV according to the assigned cohort
  Arms: IV infusion of cizutamig; SC injection of cizutamig
Other: Placebo — placebo will be dosed IV or SC according to the assigned cohort
  Arms: IV infusion of placebo; SC injection of placebo

SUMMARY:
The purpose of this study is to determine the absolute bioavailability of SC administered cizutamig in healthy adult participants.

DETAILED DESCRIPTION:
This is a randomized, double-blind, Phase 1 study designed to determine the absolute bioavailability of SC administered cizutamig in healthy adult participants. The study will enroll participants in SC and IV cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age
2. Body mass index 18-30 kg/m2 and weight 55-100 kg
3. Individuals in good health
4. Meets vaccination requirements as defined by the protocol
5. Agree to abstain from consumption of alcohol within 48-hrs of study visits
6. Agree to the use of highly effective contraception as defined by the protocol

Exclusion Criteria:

1. Active Infection
2. Inadequate clinical laboratory parameters at Screening
3. Receipt of or inability to discontinue any excluded therapies
4. Individuals who will decline blood products
5. Individuals with immediate household contacts with young children (eg, ≤ 6 years old) or immunocompromised persons
6. History of drug or alcohol abuse within last 12 months
7. Individuals who are hypersensitive to intravenous immunoglobulin (IVIg)
8. History of severe allergic or anaphylactic reactions to mAb therapy (or recombination antibody-related fusion proteins) or any constituents of study drug
9. Major surgery requiring the use of general anesthesia within 12 weeks prior to Screening or planned or expected major surgery during the study period (from Screening to the individual's last visit)
10. Blood donation or significant blood loss within 30 days prior to screening
11. Individuals considered to be part of a vulnerable population (eg, incarceration)
12. Individuals that in the opinion of the Investigator, are not suitable for participation in the trial
13. Inability to comply with protocol-mandated requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Absolute bioavailability | Baseline to 8 weeks

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events through end of study | Baseline to 8 weeks
PK parameters for cizutamig: AUC and dose-normalized AUC | Baseline to 8 weeks
PK parameters for cizutamig: Cmax and dose-normalized Cmax | Baseline to 8 Weeks
PK parameter for cizutamig: Tmax | Baseline to 8 Weeks
PK parameter for cizutamig: t½ | Baseline to 8 weeks
PK Parameters for cizutamig: CL | Baseline to 8 Weeks
  IV only
PK Parameters for cizutamig: CL/F | Baseline to 8 weeks
  SC only
Anti-drug antibodies (ADAs) | Baseline to 8 weeks
Changes in body temperature | Baseline to 8 Weeks
  oral, tympanic, or axillary
Changes in ECG parameters from baseline through end of study: QRS interval | Baseline to 8 Weeks
Changes in ECG parameters from baseline through end of study: PR interval | Baseline to 8 Weeks
Changes in ECG parameters from baseline through end of study: QTcB | Baseline to 8 Weeks
Changes in ECG parameters from baseline through end of study: QTcF | Baseline to 8 Weeks
Changes in ECG parameters from baseline through end of study: QT interval | Baseline to 8 Weeks
Changes in ECG parameters from baseline through end of study: RR | Baseline to 8 Weeks
Changes from baseline in safety laboratory assessments through end of study: serum chemistry | Baseline to 8 Weeks
PK Parameters for cizutamig: Vz | Baseline to 8 weeks
  IV only
PK Parameters for cizutamig: Vss | Baseline to 8 weeks
  IV only
PK Parameters for cizutamig: Vz/F | Baseline to 8 Weeks
  SC only
Changes in heart rate | Baseline to 8 weeks
Changes in respiratory rate | Baseline to 8 weeks
Changes in blood pressure | Baseline to 8 weeks
  systolic and diastolic
Changes in pulse oximetry | Baseline to 8 weeks
Changes from baseline in Red Blood Cell count | Baseline to 8 weeks
Changes from baseline in White Blood Cell count | Baseline to 8 weeks
Changes from baseline in Platelets | Baseline to 8 weeks
Changes from baseline in Hematocrit | Baseline to 8 weeks
Changes from baseline in Hemoglobin | Baseline to 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No